CLINICAL TRIAL: NCT03134339
Title: The Effect of Nicotine Delivery Rate on Reinforcement
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, The effect of nicotine delivery rate on reinforcement, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1609018390
Record Dates: First submitted 2017-02-06; First posted 2017-04-28 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Nicotine
Keywords: nicotine, smoking
MeSH Terms: conditions — Smoking | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: The effects of different IV nicotine delivery rates of (saline), 0.24, 0.048 and 0.024 mcg/kg/s), as a within-subject factor, on peak change in the intensity of subjective effects as measured by the DEQ, will be used as a measured of a reinforcing threshold.
Who Masked: Participant, Investigator
Masking Description: Participant and Investigator will not know nicotine dose or rate of infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- saline 0.00mcg/kg/s (Experimental): 0.00 mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine saline 0.00mcg/kg/s
- 0.24mcg/kg/s (Experimental): 0.24 mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine 0.24 mcg/kg/s
- 0.048mcg/kg/s (Experimental): 0.048 mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine 0.048 mcg/kg/s
- 0.024 mcg/kg/s (Experimental): 0.024 mcg/kg/s The day order will be randomized per day
  Interventions: Drug: Nicotine 0.024 mcg/kg/s

INTERVENTIONS:
Drug: Nicotine saline 0.00mcg/kg/s — saline 0.00mcg/kg/s
  Other Names: nicotine infusion
  Arms: saline 0.00mcg/kg/s
Drug: Nicotine 0.24 mcg/kg/s — nicotine 0.24 mcg/kg/s
  Other Names: nicotine infusion
  Arms: 0.24mcg/kg/s
Drug: Nicotine 0.048 mcg/kg/s — nicotine 0.048 mcg/kg/s
  Other Names: nicotine infusion
  Arms: 0.048mcg/kg/s
Drug: Nicotine 0.024 mcg/kg/s — nicotine 0.024 mcg/kg/s
  Other Names: nicotine infusion
  Arms: 0.024 mcg/kg/s

SUMMARY:
The dose-effect curve to estimate a threshold delivery rate for reinforcement. The project addresses the FDA Center for Tobacco Products (CTP) interest #1: Nicotine dependence threshold among youth and adults and impact of nicotine reduction on tobacco product use behavior (e.g., topography, compensation, switching, multiple use, initiation, cessation and relapse). IV nicotine, in contrast to ECs, can deliver precise, reproducible dosing, which is necessary for accurately assessing dose-response and threshold effects. The estimated threshold for reinforcement will establish a benchmark for evaluating the addictive potential of ECs and other inhaled nicotine products.

DETAILED DESCRIPTION:
A placebo-controlled study that will recruit male and female nicotine dependent smokers/EC users (n=18) to complete four separate experimental sessions. Each session will include one randomly assigned infusion that will be either saline or a single dose of nicotine (1 mg per 70 kg body weight) delivered at three different infusion rates, rapid, moderate or slow (0.24, 0.048 or 0.024 mcg per kg body weight per second). A total infusion duration of 10 min will be maintained during each session by adding saline infusions of variable duration after nicotine delivery. This will be achieved by two separate infusion pumps, one for saline and one for nicotine. For example, the rapid 0.24 mcg/kg/s condition will include a 1 min infusion of nicotine followed by a 9 min infusion of saline. The subjects will be blinded to the infusion pump procedures. The rapid delivery rate, which we have used in our prior studies, induces positive subjective drug effects and suppresses symptoms of nicotine withdrawal. The moderate delivery rate,0.048 mcg/kg/s, approximates the rate of nicotine intake encountered while smoking a typical cigarette over 5 min (4). The slowest nicotine delivery rate, 0.024mcg/kg/s, was chosen to approximate the rate of nicotine intake encountered while using a newer EC (5).

ELIGIBILITY:
Inclusion Criteria:

1. Female and male smokers that smoke ≥ 5 cigarettes per day for the past year
2. aged 18 to 30 years
3. urine cotinine levels > 100 ng/mL consistent with nicotine intake of an active smoker (23)
4. not seeking treatment at the time of the study for nicotine dependence
5. in good health as verified by medical history, screening examination, and screening laboratory tests
6. for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

1. history of major medical or psychiatric disorders that the physician investigator deems as contraindicated for the subject to be in the study
2. regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics)
3. current alcohol or substance dependence for any other recreational or prescription drugs other than nicotine
4. urine drug screening indicating recent illicit drugs use (with the exception of marijuana).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Peak Change on items of the Drug Effects Questionnaire (DEQ) | up to 60 minutes post infusion
  The peak change in the intensity of subjective effects as measured by the DEQ

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Jensen, Ph.D., Principal Investigator — Yale University; Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No